CLINICAL TRIAL: NCT06480955
Title: BOne Metastases REgistry for Patients Undergoing cryoAbLation With curatIve purpoSe
Acronym: BOREALIS
Status: Recruiting | Type: Observational
Sponsor: Cardiovascular and Interventional Radiological Society of Europe (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: BOREALIS
Record Dates: First submitted 2024-06-19; First posted 2024-06-28 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Bone Metastases
Keywords: Cryoablation Oligo-progressive disease; Bone metastases; Oligometastatic Disease; Oligo-progressive disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Full cohort: Cryoablation with curative-intent of bone metastases from oligometastatic or bone oligo-progressive disease.
  Interventions: Device: Cryoablation system

INTERVENTIONS:
Device: Cryoablation system — Any cryoablation system from Boston Scientific that has received CE Mark and/or FDA clearance for the ablation of bone malignancies.

SUMMARY:
BOREALIS is a multicentre, prospective, observational cohort study designed to investigate the effectiveness, feasibility, safety and impact on pain and quality of life of curative-intent cryoablation for the treatment of bone metastases in patients with oligometastatic or bone oligo-progressive disease.

ELIGIBILITY:
Inclusion Criteria:

* Bone metastases in patients with oligometastatic disease (<5 bone/visceral metastases) or bone oligo-progressive disease (visceral or osseous multi-metastatic disease stable under systemic treatment except 1-3 progressing bone metastases) from solid tumours;
* Number of target lesions ≤ 3
* Size of target lesion(s) < 5 cm (largest diameter);
* Referral to local ablative treatment by multidisciplinary tumour board (MDTB);
* Treatment by percutaneous cryoablation with curative intent (i.e., complete tumour destruction) assessed as technically feasible by the IR in charge;
* Procedure performed with a cryoablation system from Boston Scientific.

Exclusion Criteria:

* < 18 years old;
* Incapacity or refusal to give informed consent;
* Ongoing pregnancy;
* Health status not compatible with the minimum meaningful follow-up period (i.e., 12 months):

  * Karnofsky Performance Scale < 60%, or
  * Bone metastases originating from rapidly evolving tumour histologies not allowing reasonable life expectancy of at least 12 months, or
  * Life expectancy < 12 months
* Infection of treatment site or systemic infection;
* Uncorrectable coagulopathy;
* Haematological disease (including multiple myeloma and plasmacytoma);
* Concomitant radiation therapy or radiation therapy within 12 weeks before the planned cryoablation procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bone metastases from oligometastatic or bone oligo-progressing disease from solid tumours treated with curative-intent cryoablation may participate in BOREALIS. Patients from vulnerable populations (e.g., minors, pregnant women, incapacitated or unconscious individuals) shall not be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Local progression-free survival rate | 12 months
  On a per lesion basis, proportion of target lesions free from local tumour progression using the Kaplan Meier estimate

SECONDARY OUTCOMES:
Technical feasibility | Periprocedurally
  Adherence to a comprehensive SOC treatment protocol that includes i) peri-operative biopsy if indicated, ii) cryoablation, and iii) bone consolidation through osteoplasty or osteosynthesis if biomechanically indicated
Adverse events | Through study completion
  Incidence and severity of adverse events graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Complete local tumour response | 12 months
  On a per lesion basis, proportion of target lesions with complete response status
Fracture-free survival | End of study
  On a per lesion basis,time between cryoablation and fracture at treated site
Fracture-free survival rate | Until the end of the follow-up period (1 year)
  On a per lesion basis, proportion of target lesion(s) free from fracture
Bone-disease progression-free survival | Until the end of the follow-up period (1 year)
  Time between cryoablation and progression in the bone (incl. new lesions)
Extraosseous disease progression-free survival | Until the end of the follow-up period (1 year)
  Time between cryoablation and extra-osseous progression (incl. new lesions)
Overall progression-free survival | Until the end of the follow-up period (1 year)
  Time between cryoablation and any progression (incl. new lesions) or death
Overall survival | Until the end of the follow-up period (1 year)
  Time between cryoablation and death
Systemic therapy-free survival | Until the end of the follow-up period (1 year)
  Time between cryoablation and the next systemic treatment (excluding any adjuvant treatment that was part of the patient's treatment plan)
Impact on patient pain | 1, 3, 6, 12 months
  Patient-reported pain assessment using the Brief Pain Inventory - short form
Impact on patient quality of life | 1, 3, 6, 12 months
  Patient-reported quality of life assessment using the EORTC QLQ-C30 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Roberto L Cazzato, Dr, Study Chair — Strasbourg University Hospitals, Strasbourg, France
Locations (5):
- France (3):
  - Institute Bergonié, Bordeaux
  - CHRU de Strasbourg, Strasbourg
  - Institut Gustave Roussy, Villejuif
- Hospital Universitario y Politécnico La Fe, Valencia, Spain
- CHUV-Lausanne University Hospital, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No